CLINICAL TRIAL: NCT02731742
Title: A Phase 1/1b Trial of MK-1966 in Combination With SD-101 in Subjects With Advanced Malignancies
Brief Title: Dose Evaluation of MK-1966 in Combination With SD-101 in Participants With Advanced Malignancies (MK-1966-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1966-001; MK-1966-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-04-04; First posted 2016-04-07 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-09

CONDITIONS: Neoplasms, Advanced
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose A MK-1966 + Dose A SD-101 (Experimental): Participants received a combination of MK-1966 (Days 1 and 21) and SD-101 (Days 1, 8, 15 and Day 22) in Part A of the study (approximately 21 days). Participants were to continue in one of two expansion cohorts (Part B or C) and receive up to 8 cycles of treatment (approximately 24 weeks). Each cycle was 21 days.
  Interventions: Biological: MK-1966; Drug: SD-101
- Dose A MK-1966 + Dose B SD-101 (Experimental): Participants received a combination of MK-1966 (Days 1 and 21) and SD-101 (Days 1, 8, 15 and Day 22) in Part A of the study (approximately 21 days). Participants were to continue in one of two expansion cohorts (Part B or C) and receive up to 8 cycles of treatment (approximately 24 weeks). Each cycle was 21 days.
  Interventions: Biological: MK-1966; Drug: SD-101
- Dose B MK-1966 + Dose B SD-101 (Experimental): Participants received a combination of MK-1966 (Days 1 and 21) and SD-101 (Days 1, 8, 15 and Day 22) in Part A of the study (approximately 21 days). Participants were to continue in one of two expansion cohorts (Part B or C) and receive up to 8 cycles of treatment (approximately 24 weeks). Each cycle was 21 days.
  Interventions: Biological: MK-1966; Drug: SD-101
- Dose C MK-1966 + Dose B SD-101 (Experimental): Participants received a combination of MK-1966 (Days 1 and 21) and SD-101 (Days 1, 8, 15 and Day 22) in Part A of the study (approximately 21 days). Participants were to continue in one of two expansion cohorts (Part B or C) and receive up to 8 cycles of treatment (approximately 24 weeks). Each cycle was 21 days.
  Interventions: Biological: MK-1966; Drug: SD-101
- Part B Expansion Cohort (Experimental): Participants were to receive the MTD/MAD of MK-1966 and SD-101 established in Part A for up to 7 additional treatment cycles with MK-1966 and up to 6 additional treatment cycles with SD-101. Each cycle was to be 21 days.
  Interventions: Biological: MK-1966; Drug: SD-101
- Part C Expansion Cohort (Experimental): Participants were to receive the MTD/MAD of MK-1966 and SD-101 established in Part A for up to 7 additional treatment cycles with MK-1966 and 6 additional treatment cycles with SD-101. Each cycle was to be 21 days.
  Interventions: Biological: MK-1966; Drug: SD-101

INTERVENTIONS:
Biological: MK-1966 — MK-1966 administered as an intravenous (IV) infusion
Drug: SD-101 — SD-101 administered as an intratumoral (IT) injection

SUMMARY:
This was a non-randomized, open-label study of MK-1966 used in combination with SD-101 in the treatment of advanced malignancies. The study included an initial Dose Evaluation phase (Part A) to determine the maximum tolerated dose (MTD)/maximum administered dose (MAD) by evaluating Dose Limiting Toxicities (DLTs) of four dose combinations of MK-1966 and SD-101. Following determination of the MTD/MAD, approximately 20 participants each were to be enrolled in two expansion cohorts (Parts B or C) to confirm/refine the MTD/MAD. The study was terminated by the Sponsor before enrollment into Part A concluded and before enrollment into Parts B and C began.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced malignancy that has progressed after standard-of-care therapy/treatments and there is no available therapy likely to convey clinical benefit
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Has a life expectancy ≥ 6 months
* Female participants must not be pregnant (negative urine or serum human chorionic gonadotropin test at screening and again within 72 hours prior to receiving the first dose of study therapy)
* Female and male participants of reproductive potential must agree to use adequate contraception during the course of the study through 120 days after study the last dose of study therapy
* Has ability to submit archived or fresh tumor sample during the screening period

Exclusion Criteria:

* Has had chemotherapy, radiation, or biological cancer therapy within 4 weeks prior to the first dose of study therapy, or who has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better from the adverse events due to cancer therapeutics administered more than 4 weeks earlier
* Has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days of study start
* Is expected to require any other form of antineoplastic therapy while on study
* Is on chronic systemic steroid therapy in excess of replacement doses, or on any other form of immunosuppressive medication
* Has a history of a malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 5 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has had a severe hypersensitivity reaction to treatment with another monoclonal antibody
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has an active infection requiring therapy
* Has active, current pneumonitis, or a history of (non-infectious) pneumonitis that required steroids
* Has had a prior stem cell or bone marrow transplant
* Is positive for Human Immunodeficiency Virus (HIV) and/or Hepatitis B or C
* Has known psychiatric disorder that would interfere with fulfilling the requirements of the study
* Is a regular user of any illicit drugs or had a recent history of substance abuse
* Has symptomatic ascites or pleural effusion
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study
* Has clinically significant heart disease that affects normal activities
* Has had major surgery (requiring at least a 3 day hospital stay) in the past 28 days
* Has received a live vaccine within 30 days prior to first dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated prior to completion of Part A enrollment and prior to initiation of Parts B or C enrollment. This results disclosure is for Part A only.
Groups:
- MK-1966 70 mg+SD-101 1 mg: Participants received a combination of MK-1966 70 mg intravenously (IV) (on Day 1 of each 3-week cycle for up to 8 cycles) and SD-101 1 mg intratumorally (IT) (on Days 1, 8 and 15 of Cycle 1, and then on Day 1 of up to 7 additional 3-week cycles) in Part A of the study. Participants were then to continue in one of two expansion cohorts (Part B or C) and were to receive up to 8 cycles of treatment on Day 1 of each 3-week cycle (approximately 24 weeks), but the study was terminated by the Sponsor prior to completion of Part A enrollment and prior to initiation of Parts B or C enrollment.
- MK-1966 70 mg+SD-101 4 mg: Participants received a combination of MK-1966 70 mg IV (on Day 1 of each 3-week cycle for up to 8 cycles) and SD-101 4 mg IT (on Days 1, 8 and 15 of Cycle 1, and then on Day 1 of up to 7 additional 3-week cycles) in Part A of the study. Participants were then to continue in one of two expansion cohorts (Part B or C) and were to receive up to 8 cycles of treatment on Day 1 of each 3-week cycle (approximately 24 weeks), but the study was terminated by the Sponsor prior to completion of Part A enrollment and prior to initiation of Parts B or C enrollment.
- MK-1966 210 mg+SD-101 4 mg: Participants received a combination of MK-1966 210 mg IV (on Day 1 of each 3-week cycle for up to 8 cycles) and SD-101 4 mg IT (on Days 1, 8 and 15 of Cycle 1, and then on Day 1 of up to 7 additional 3-week cycles) in Part A of the study. Participants were then to continue in one of two expansion cohorts (Part B or C) and were to receive up to 8 cycles of treatment on Day 1 of each 3-week cycle (approximately 24 weeks), but the study was terminated by the Sponsor prior to completion of Part A enrollment and prior to initiation of Parts B or C enrollment.
- MK-1966 700 mg+SD-101 4 mg: Participants received a combination of MK-1966 700 mg IV (on Day 1 of each 3-week cycle for up to 8 cycles) and SD-101 4 mg IT (on Days 1, 8 and 15 of Cycle 1, and then on Day 1 of up to 7 additional 3-week cycles) in Part A of the study. Participants were to continue in one of two expansion cohorts (Part B or C) and were to receive up to 8 cycles of treatment on Day 1 of each 3-week cycle (approximately 24 weeks), but the study was terminated by the Sponsor prior to completion of Part A enrollment and prior to initiation of Parts B or C enrollment.
Period: Overall Study
Arm/Group | MK-1966 70 mg+SD-101 1 mg | MK-1966 70 mg+SD-101 4 mg | MK-1966 210 mg+SD-101 4 mg | MK-1966 700 mg+SD-101 4 mg
Started | 3 | 3 | 6 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 2
Not completed — Death | 1 | 2 | 5 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1966 70 mg+SD-101 1 mg | MK-1966 70 mg+SD-101 4 mg | MK-1966 210 mg+SD-101 4 mg | MK-1966 700 mg+SD-101 4 mg | Total
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (1.5) | 63.0 (6.9) | 63.7 (6.8) | 50.5 (2.1) | 61.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3 | 1 | 7
  Male | 0 | 3 | 3 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 2 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Dose Limiting Toxicity (DLT)
Description: The occurrence of any of the following toxicities during Cycle 1 (Days 1-21), if assessed by the Investigator to be possibly, probably or definitely related to MK-1966 or SD-101, was considered a DLT:
  1. Grade (Gr) 4 non-hematologic toxicity;
  2. Gr 4 hematologic toxicity lasting >7 days, except thrombocytopenia: *Gr 4 thrombocytopenia of any duration; *Gr 3 thrombocytopenia if associated with bleeding;
  3. Gr 3 non-hematologic toxicity lasting >3 days despite optimal supportive care;
  4. Any Gr 3 or Gr 4 non-hematologic laboratory abnormality, if: medical intervention is required OR abnormality leads to hospitalization OR abnormality persists for >1 week;
  5. Febrile neutropenia Gr 3 or Gr 4;
  6. Any drug-related AE which caused participant to discontinue study drug during Cycle 1
  7. Gr 5 toxicity; or
  8. Delay in initiation of Cycle 2 for >2 weeks due to study drug-related toxicity. The percentage of participants who experienced a DLT during Cycle 1 is presented.
Time Frame: From time of first dose of study drug to the end of Cycle 1. Each cycle was 21 days. (Up to 21 days)
Population: The DLT evaluable population consisted of all participants who completed study drug in Cycle 1 or discontinued study drug during Cycle 1 due to a DLT.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-1966 70 mg+SD-101 1 mg | MK-1966 70 mg+SD-101 4 mg | MK-1966 210 mg+SD-101 4 mg | MK-1966 700 mg+SD-101 4 mg
Number analyzed (Participants) | 3 | 3 | 5 | 2
Percentage of Participants | 0.0 [0.0 to 33.1] | 0.0 [0.0 to 33.1] | 20.0 [5.1 to 44.8] | 0.0 [0.0 to 41.5]

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study drug, was also an AE. The number of participants who experienced as AE is presented.
Time Frame: From first dose of study drug through 90 days after last dose of study drug (Up to approximately 22 weeks)
Population: The safety analysis population consisted of all participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1966 70 mg+SD-101 1 mg | MK-1966 70 mg+SD-101 4 mg | MK-1966 210 mg+SD-101 4 mg | MK-1966 700 mg+SD-101 4 mg
Number analyzed (Participants) | 3 | 3 | 6 | 2
Participants | 3 | 3 | 6 | 2

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to AEs
Description: The number of participants who discontinued study drug due to an AE is presented.
Time Frame: From first dose of study drug up to last dose of study drug (Up to approximately 9 weeks)
Population: The safety analysis population consisted of all participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1966 70 mg+SD-101 1 mg | MK-1966 70 mg+SD-101 4 mg | MK-1966 210 mg+SD-101 4 mg | MK-1966 700 mg+SD-101 4 mg
Number analyzed (Participants) | 3 | 3 | 6 | 2
Participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 90 days after last dose of study drug (Up to approximately 22 weeks)
Description: The safety analysis population consisted of all participants who received ≥1 dose of study drug.
  Per protocol, progression of cancer under study was not considered an AE unless related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | MK-1966 70 mg+SD-101 1 mg | MK-1966 70 mg+SD-101 4 mg | MK-1966 210 mg+SD-101 4 mg | MK-1966 700 mg+SD-101 4 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 5/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 3/6 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1966 70 mg+SD-101 1 mg (N=3) | MK-1966 70 mg+SD-101 4 mg (N=3) | MK-1966 210 mg+SD-101 4 mg (N=6) | MK-1966 700 mg+SD-101 4 mg (N=2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1966 70 mg+SD-101 1 mg (N=3) | MK-1966 70 mg+SD-101 4 mg (N=3) | MK-1966 210 mg+SD-101 4 mg (N=6) | MK-1966 700 mg+SD-101 4 mg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (6) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (3) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 3 (3) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervigilance (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02731742/Prot_SAP_000.pdf